CLINICAL TRIAL: NCT05356858
Title: An Open Label Trial Evaluating the Efficacy and Safety of Bruton's Tyrosine Kinase (BTK) Inhibitor Zanubrutinib in Adult Patients With Neuromyelitis Optical Spectrum Disorders (NMOSDs)
Brief Title: An Open Label Study of the Effects and Safety of Zanubrutinib in NMOSDs Adult Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-2005-IIT
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-04

CONDITIONS: Neuromyelitis Optica
Keywords: NMOSD; BTK inhibitor,; zanubrutinib
MeSH Terms: conditions — Neuromyelitis Optica | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zanubrutinib (Experimental): zanubrutinib orally, 80mg bid for 1 year
  Interventions: Drug: zanubrutinib

INTERVENTIONS:
Drug: zanubrutinib — zanubrutinib orally, 80mg bid for 1 year

SUMMARY:
This is an open-label study, to evaluate the efficacy and safety of a BTK inhibitor zanubrutinib in participants with NMOSDs.

DETAILED DESCRIPTION:
This is an open, single-center clinical study to evaluate the efficacy and safety of Zanubrutinib in the treatment of recurrent neuromyelitis optica spectrum disease. Patients were required to be diagnosed with neuromyelitis optic spectrum disease according to the NMOSD diagnostic criteria established by the international NMO Diagnostic Group (IPND) in 2015, and to have had at least two relapses (including first episode) within two years while at least one relapse occurring within the 12 months prior to screening. The AQP4 antibody must be positive during screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the NMOSD diagnostic criteria set by the international NMO Diagnostic Group (IPND) in 2015.
* Serum AQP4-IgG positive.
* Clinical evidence of at least 2 documented relapse (including first attack) in the last 2 years, with at least 1 relapse within 12 months prior to screening.
* Extended Disability Status Scale (EDSS) score ≤7.5 at screening.
* Age 18 to 75 years inclusive, weight at least 35 kg at the time of informed consent.
* If the patients were using the following baseline treatment for relapse prevention, they must be treated at a steady dose for at least 4 weeks prior to enrollment:

  * Azathioprine, metecophenol ester and other immunosuppressive agents
  * Oral corticosteroid (≦30mg/ day prednisone tablet or equivalent dose of other hormones)
* (patients or their legal representatives) can provide written informed consent indicating that they understand and agree to comply with the requirements of the study protocol.

Exclusion Criteria:

* Continuous treatment with strong or moderate CYP3A inhibitors or inducers is required during the study period. Patients were excluded if they had taken a potent or moderate CYP3A inhibitor or inducer within 7 days prior to administration of the study drug (or had stopped taking these drugs for less than 5 half-lives).
* Previously treated with BTK inhibitors (e.g., ibrutinib).
* Allergic to the study drug or any of the ingredient.
* Desease relaps (including first episode) within the previous 30 days.
* Pregnancy or lactation.
* Previous or current malignancy, except locally recurrent cancers that have received radical treatment (e.g. excised basal or squamous cell skin cancer, cervical or breast cancer in situ).
* Currently central nervous system (CNS) disease that may affect the evaluation of NMOSD.
* Serious and uncontrolled conditions considered by the investigator that could affect safety, compliance and endpoint evaluation, or need for use of a drug not permitted in the protocol.
* Disease that could affected drug absorption, distribution, metabolism, and excretion determined by the investigator.
* Any major clinical infection lead to hospitalization or parenteral antibiotic treatment within 1 month prior to screening; Or other infections that may be aggravated due to the study determined by the investigator.
* Active, latent or undertreated mycobacterium tuberculosis (TB) infection
* Known primary immunodeficiency or underlying disease such as human immunodeficiency virus (HIV) infection.
* Hepatitis B or C virus infection by serological test.
* Received B-cell targeted therapy (e.g. Rituximab) within 6 months prior to the initial administration of the study drug.
* Received biologics such as tozizumab within 12 weeks prior to initial administration of the study drug.
* Received live attenuated vaccine during the screening and study periods, or any live virus vaccine within 8 weeks prior to initial administration.
* Abnormal and clinically significant in ECG examination during screening.
* Uncontrolled hypertension (SBP>160 mmHg or DBP ≥ 95 mmHg)
* Grade 3 or 4 heart Failure, (NYHA scale).
* Severe liver insufficiency (Child-pugh C).
* Aspartate aminotransferase (AST)>3 times the upper limit of normal (ULN) and/or alanine aminotransferase (ALT)>3ULN and/or bilirubin >2ULN.
* Estimated creatinine clearance <30 mL/min or requiring dialysis.
* Inability to receive MRI scans
* A history of clinically significant CNS trauma
* Received experimental drug or other experimental treatment within 4 weeks prior to screening or during 5 pharmacokinetic half-lives or duration of biological effects, whichever is longer.
* Participate in another clinical study.
* Accept any of the following:

  * BCG vaccination within 1 year prior to screening.
  * Prior bone marrow transplant, hematopoietic stem cell transplant, or systemic radiation therapy.
  * Received intravenous gamma globulin within 30 days prior to screening.
  * Plasmapheresis or leukocyte separation within 90 days prior to screening
* Abnormal white blood cell count, neutrophil count, lymphocyte count, or platelet count during the screening and were considered unsuitable for study by investigator
* Inability to swallow capsules or medical conditions that significantly affect gastrointestinal function
* A history of severe hemorrhagic disorders such as hemophilia A, hemophilia B, von willebrand disease, or a history of spontaneous bleeding requiring blood transfusion or other medical intervention.
* History of stroke or intracranial hemorrhage within 6 months prior to screening
* Current alcohol, drug or chemical abuse, or history of such abuse within 1 year prior to screening.
* Anticoagulants or a combination of anticoagulants and antiplatelet agents is ongoing or planned.
* Any other circumstances in which the investigator or sponsor considers the patient unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Relapse-free rate at week 48 | up to week 48
  Proportion of subjects who are relapse-free at week 48

SECONDARY OUTCOMES:
Changes in the expanded disability status scale (EDSS) score from baseline at week 12,24,36 and 48 | up to week12,24,36 and 48
  EDSS is an ordered scale with values ranging from 0 points (normal neurological examination) to 10 points (death) in increments of 0.5 points. Higher scores indicate increased disability, and negative changes from baseline indicate improvement
Changes in visual acuity at week 12, 24,36 and 48 from baseline | up to week12,24,36 and 48
  Changes in visual acuity at week 12, 24,36 and 48 from baseline
Changes in the MOS item short from health survey (SF-36) score at week 12, 24,36 and 48 from baseline | up to week12,24,36 and 48
  The SF-36 is a multi-purpose, concise 36-question health survey scale. It contains 8 dimensions,The eight dimensions were converted to a scale of 0-100, with a higher score indicating a better quality of life. Positive change from baseline indicates improvement.
Changes in Serum AQP4-IgG titer at week 12, 24,36 and 48 from baseline | up to week12,24,36 and 48
  Changes in Serum AQP4-IgG titer at week 12, 24,36 and 48 from baseline
Changes in Peripheral blood lymphocyte subset at week 12, 24,36 and 48 from baseline | up to week12,24,36 and 48
  Changes in Peripheral blood lymphocyte subset at week 12, 24,36 and 48 from baseline
Plasma concentraion of zanubrutinib | up to week 48
  Concentraion of zanubrutinib in peripheral blood plasma
Number of participants with all grade Adverse Events, Serious Adverse Events and who discontinued study therapy due to AEs | up to week 48
  Evaluate Number of participants with all grade Adverse Events and Serious Adverse Events determined by NCI-CTCAE V5.0，and tolerance base on percentage of patients who discontinued study therapy due to AEs

OTHER OUTCOMES:
Concentraion of zanubrutinib in Cerebrospinal fluid at week 12 | up to week 12
  Concentraion of zanubrutinib in Cerebrospinal fluid at week 12
BTK accupancy of peripheral blood mononuclear cells | up to week 48
  BTK accupancy of peripheral blood mononuclear cells in NMOSD patients before zebutinib administration, 4-6h after zebutinib administration, and at weeks 12 and 48.

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, MD, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- XuanWu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No